CLINICAL TRIAL: NCT01432431
Title: Archstone Spiritual Care Demonstration Project: Outcomes for Patients, Families, and Staff
Brief Title: Spiritual Care in Improving Quality of Life of Patients, Caregivers, and Hospital Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11110; NCI-2011-02730 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Spiritual Therapies; Counseling; Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (spiritual care) (Experimental): See Detailed Description.
  Interventions: Procedure: spiritual therapy; Other: questionnaire administration; Other: survey administration; Other: counseling intervention; Other: psychosocial support for caregiver; Procedure: psychosocial assessment and care

INTERVENTIONS:
Procedure: spiritual therapy — Undergo palliative spiritual care
  Other Names: spirituality
Other: questionnaire administration — Ancillary studies
Other: survey administration — Ancillary studies
Other: counseling intervention — Undergo palliative spiritual care
  Other Names: counseling and communications studies
Other: psychosocial support for caregiver — Undergo palliative spiritual care
Procedure: psychosocial assessment and care — Undergo palliative spiritual care
  Other Names: psychosocial assessment; psychosocial assessment/care; psychosocial care; psychosocial care/assessment; psychosocial studies

SUMMARY:
This clinical trial studies spiritual care in improving quality of life of patients, caregivers, and hospital staff. Spiritual care may help understand the impact cancer and its treatment has on patients, caregivers and hospital staff.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To improve the quality of spiritual care provided by palliative care teams. II. To measure the effectiveness of integrating spiritual care recommendations in palliative care at City of Hope (COH) and the impact it has on cancer patients, families, and hospital staff.

OUTLINE:

The expanded psychosocial/spiritual assessment administered by social workers includes a spiritual history and a spiritual needs screening. Social worker knowledge and competence is surveyed at baseline, immediately after the course, and after a bedside chaplain-mentoring process. Inpatient cancer patients' and their caregivers' perceptions about spiritual care is surveyed at baseline prior to the social work curriculum and after the course has been completed and the new psychosocial/spiritual assessment has been implemented. Data collected from patients, family members, and staff includes number of unduplicated palliative care patients screened for spiritual concerns, spiritual history, number and type of spiritual issues, number of referrals to the chaplain, number seen by the chaplain, number of unduplicated palliative care patients with documented spiritual care plan, number of staff development sessions offered and topics, attendance per topic, advance directives, and referrals to hospice.

ELIGIBILITY:
Inclusion Criteria:

* Admitted during the study quarter
* Admitted >= 5 days
* English speaking
* Alert and able to answer questions

Exclusion Criteria:

* Non-cancer diagnosis
* Previously accrued to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change over time in number of unduplicated palliative care patients screened for spiritual concerns and spiritual history | At baseline and quarterly for one year
  Nonparametric Mann-Whitney University test will be used to test for differences between cohorts of patients and of families at the two different measurement points. The Wilcoxon paired nonparametric test will be used to test for change over time for staff survey results.
Change over time in number and type of spiritual issues | At baseline and quarterly for one year
  Nonparametric Mann-Whitney University test will be used to test for differences between cohorts of patients and of families at the two different measurement points. The Wilcoxon paired nonparametric test will be used to test for change over time for staff survey results.
Change over time in number of referrals to the chaplain and number seen by the chaplain | At baseline and quarterly for one year
  Nonparametric Mann-Whitney University test will be used to test for differences between cohorts of patients and of families at the two different measurement points. The Wilcoxon paired nonparametric test will be used to test for change over time for staff survey results.
Change over time in number of unduplicated palliative care patients with documented spiritual care plan | At baseline and quarterly for one year
  Nonparametric Mann-Whitney University test will be used to test for differences between cohorts of patients and of families at the two different measurement points. The Wilcoxon paired nonparametric test will be used to test for change over time for staff survey results.
Change over time in number of staff development sessions offered and topics, attendance per topic, advance directives, and referrals to hospice | At baseline and quarterly for one year
  Nonparametric Mann-Whitney University test will be used to test for differences between cohorts of patients and of families at the two different measurement points. The Wilcoxon paired nonparametric test will be used to test for change over time for staff survey results.
Identification of common themes and patterns that answer the key evaluation questions | At baseline and quarterly for one year
  Analyzed using Atlas.ti. coding and analysis. Qualitative data, e.g., open ended questions, included narrative responses by staff summarized for reporting purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Thomas, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States